CLINICAL TRIAL: NCT04158115
Title: Comparison Between Segmental Mobilization And Entire Spine Mobilization In Lumbar Spondylosis
Brief Title: Segmental Mobilization vs Entire Spine Mobilization In Lumbar Spondylosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sadaf nisar REC/00343
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Spondylosis Lumbar
Keywords: Lumber Spondylosis; Segmental Mobilization; Spine Mobilization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Entire Spinal Mobilization (Experimental): Entire Spinal Mobilization( All spinal segment from Co-C1to L5-S1 Moist heat. Soft tissue Mobilization Exercises. (Knee to chest, Bridging. Hamstrings Stretching, TA stretching)
  Interventions: Other: Entire Spine Mobilization
- Segmental Mobilization (Active Comparator): Segmental Mobilization. (All lumbar segment from L1-L2 to L5-S1) Moist heat. Soft tissue Mobilization Exercises (Knee to chest, Bridging. Hamstrings Stretching, TA stretching)
  Interventions: Other: Segmental Mobilization

INTERVENTIONS:
Other: Entire Spine Mobilization — 8 sessions of Following: -Entire Spinal Mobilization of all spinal segment from C0 to C1 to L5 to S1 (10 reps × 3 sets), - Moist heat: 10 to 15 minutes, - Soft tissue Mobilization, - Exercises : (Knee to chest, Bridging. Hamstrings Stretching, TA stretching)
  Arms: Entire Spinal Mobilization
Other: Segmental Mobilization — 8 sessions of following -Segmental Mobilization: All lumbar segment from L1 to L2 to L5 to S1 (10 reps × 3 sets) - Moist heat: (10 to 15 minutes), -Soft tissue Mobilization
  - Exercises: (Knee to chest, Bridging. Hamstrings Stretching, TA stretching)
  Arms: Segmental Mobilization

SUMMARY:
This study will compare the effect of segmental spine mobilization and entire spine mobilization in the patients with lumber spondylosis.

There will be two groups ; experimental and control. Half of study group will receive segmental mobilization along with conventional treatment such as moist heat , soft tissue mobilization and traditional stretching exercises and half of study group will receive entire spine mobilization along with the same conventional treatment given to other group.

DETAILED DESCRIPTION:
This is a randomized controlled trial which is being conducted in Pakistan Railway hospital enrolled total 40 participants diagnosed with lumbar spondylosis who fulfilled the inclusion criteria through sealed envelope method using purposive sampling technique into two groups I-e experimental (n=21) and control group(n=19).The treatment protocol administered to experimental group was Maitland entire spine mobilization along with other conventional treatments such as hot pack, soft tissue mobilization.

and home-based exercises (Bridging, knee to chest, Hamstrings stretching and TA stretching). While the control group received segmental spine mobilization along with same conventional treatment as mentioned above for 8 sessions. Physical therapy along with pharmaceutical management is effective in improving pain on NPRS, ODI values in patients with lumbar stenosis. Based on evidence that manual therapy interventions when used in combination with exercise therapy in clinical practice has beneficial effect in the treatment of degenerated lumbar spinal stenosis.

effects of 'specific segmental level 'spinal joint mobilization techniques in creating positive outcomes on pain NPRS measures and range of motion concluded that a single session of segmental joint mobilization can lead to pain reduction at both rest and with most painful offending movement.

Manual therapy approaches such as Maitland mobilizations are more productive in the management of chronic low back pain, quality of function and lumbar spine range of motion in patients of lumbar spondylosis than traditional physical therapy interventions such as muscle stretching and spinal traction.

Osteophytes were the most numerous radiographic feature detected in patients with lumbar spondylosis, with greater occurrence in men. Intervertebral disc space narrowing was more prevalent in women than men. Both distinctive radiographic features presence increased with increasing age. Disc space reduction seemed more strongly related with chronic low back pain than osteophytosis, especially in men and disc space narrowing at 2 or more segments appeared more powerfully associated with low back pain than disc space reduction at only 1 intervertebral segment.

Maitland posteroanterior spinal mobilizations are performed by a therapist on symptomatic segments after assessment compared with mobilization treatment given on any random spinal segment in patients suffering with chronic low back pain. The results were greater degree of immediate reduction of pain in patients receiving posteroanterior mobilization on symptomatic segment rather than any random segments in offending movement direction.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar spondylosis.
* Limited ROM (at least two)
* Symptoms more than month

Exclusion Criteria:

* Spinal stenosis.
* Osteoporosis in X-ray.
* Significant Trauma/Fracture (with in last 06 month)
* Spondylolysis.
* Inflammatory arthritis.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 8th day
  Oswestry disability index is basically a tool established by Jeremy Fairbank et al to measure functional outcome and quality of life of persons suffering from low back pain. It consists of total of 10 questions, Every question sores from 0-5 containing 6 questions, which constitutes total of 60 marks for 10 questions. By increasing the value of ODI degree of disability increases. If the percentage fall in 0-20% it indicates minimal disability.21-40% indicates moderately disabled persons, 41 -60% demonstrates severely disabled persons. 61- 80% showed crippled and above 80 are bed bound or psychologically ill patient. Percentages were taken on 1st, 4th and 8th visits to determine the quality of life of patients.
Numeric Pain Rating Scale (NPRS) | 8th Day
  NPRS values was taken as baseline assessment on 1st visit and post intervention assessment after 1st session. Then again, readings were taken on 4th visit. And final reading was taken on 8th visit for both back and legs.
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme. Scores range from 0-10 points, with higher scores indicating greater pain intensity.
Spine goniometry | 8th day
  We also measured lumbar flexion, extension, right and left side bending at both baseline and end results after 1st 4th and 8th session of treatment in both the control and experimental groups.

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Ghafoor Sajjad, Phd*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International university, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reiman MP, Harris JY, Cleland JA. Manual therapy interventions for patients with lumbar spinal stenosis: a systematic review. InDatabase of Abstracts of Reviews of Effects (DARE): Quality-assessed Reviews [Internet] 2009. Centre for Reviews and Dissemination (UK).
- [Background] Slaven EJ, Goode AP, Coronado RA, Poole C, Hegedus EJ. The relative effectiveness of segment specific level and non-specific level spinal joint mobilization on pain and range of motion: results of a systematic review and meta-analysis. J Man Manip Ther. 2013 Feb;21(1):7-17. doi: 10.1179/2042618612Y.0000000016. PMID 24421608
- [Background] Sharma A, Alahmari K, Ahmed I. Efficacy of Manual Therapy versus Conventional Physical Therapy in Chronic Low Back Pain Due to Lumbar Spondylosis. A Pilot Study. Med Sci (Basel). 2015 Jun 26;3(3):55-63. doi: 10.3390/medsci3030055. PMID 29083391
- [Background] Osama, Muhammad & Malik, Reem & Ahmad, Shakeel. (2017). Effects of facet joint mobilization in patients with straightening of the cervical spine: A pilot study. 10.13140/RG.2.2.15585.10083.